CLINICAL TRIAL: NCT02336815
Title: A Phase 2b, Open-Label, Single-Arm Study of Selinexor (KPT-330) Plus Low-Dose Dexamethasone (Sd) in Patients With Multiple Myeloma Previously Treated With Lenalidomide, Pomalidomide, Bortezomib, Carfilzomib, and an Anti-CD38 Monoclonal Antibody (mAb) Daratumumab, and Refractory to Prior Treatment With Glucocorticoids, an Immunomodulatory Agent, a Proteasome Inhibitor, and an the Anti-CD38 mAb Daratumumab
Brief Title: Selinexor Treatment of Refractory Myeloma
Acronym: STORM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-012
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Karyopharm; KPT-330; Selinexor; Refractory; Bortezomib; Carfilzomib; Lenalidomide; Pomalidomide; Dexamethasone; STORM; Daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 (Experimental): Participants with quad-exposed, double-class-refractory (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, but not an anti-CD38 mab) and penta-exposed, triple-class-refractory multiple myeloma (MM) (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, and daratumumab, and refractory to prior treatment with glucocorticoids, an immunomodulatory agent (IMiD), a proteasome inhibitor (PI), and the anti-CD38 mAb daratumumab) received, two dosing schedules (1) Selinexor 80 milligrams (mg) plus low-dose dexamethasone 20 mg (Sd) twice-weekly on Days 1 and 3 for 3 weeks of each 4-week cycle (2) Selinexor 80 mg plus low-dose dexamethasone 20 mg (Sd) twice-weekly continuously in 4-week cycles; until disease progression, death, or unacceptable toxicity (maximum duration of approximately 13 months).
  Interventions: Drug: Selinexor; Drug: Dexamethasone
- Part 2 (Experimental): Participants who previously had received more than 3 anti-MM regimens and had penta-exposed, triple class-refractory MM (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, and daratumumab, and refractory to prior treatment with glucocorticoids, an IMiD, a PI, and the anti-CD38 mAb daratumumab) received, Selinexor 80 mg post oral (PO) plus low-dose dexamethasone 20 mg Sd twice-weekly on Days 1 and 3 until disease progression, death, or unacceptable toxicity (maximum duration of approximately 17 months).
  Interventions: Drug: Selinexor; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Fixed oral dose of 80 mg twice weekly (e.g., Monday and Wednesday or Tuesday and Thursday, etc.)
  Other Names: KPT-330
Drug: Dexamethasone — 20 mg was given with each dose of Selinexor.

SUMMARY:
This is a Phase 2b, single-arm, open-label, multicenter study of selinexor 80 mg plus dexamethasone 20 mg (Sd) dosed twice weekly in four-week cycles, in patients with penta-refractory MM (Parts 1 and 2) or quad refractory MM (Part 1 only).

DETAILED DESCRIPTION:
This is a Phase 2b, single-arm, open-label, multicenter study of selinexor 80 mg plus dexamethasone 20 mg (Sd), both dosed twice weekly in each four-week cycle, in patients with MM previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, and daratumumab and refractory to prior treatment with glucocorticoids, an immunomodulatory agent (IMiD), a proteasome inhibitor (PI), and daratumumab.

This study consists of two parts:

* Part 1 enrolled patients with both quad-refractory MM and penta-refractory MM.
* Part 2 will enroll patients with penta-refractory MM only.

ELIGIBILITY:
Inclusion Criteria:

Measurable MM based on modified IMWG guidelines. Defined by at least one of the following:

1. Serum M-protein ≥ 0.5 g/dL by serum electrophoresis (SPEP) or for IgA myeloma, by quantitative IgA
2. Urinary M-protein excretion ≥ 200 mg/24 hours
3. Free Light Chain (FLC) ≥ 100 mg/L, provided that the FLC ratio is abnormal
4. If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative Ig levels by nephelometry or turbidimetry are acceptable

   * Must have previously received ≥ 3 anti-MM regimens including: an alkylating agent, lenalidomide, pomalidomide, bortezomib, carfilzomib, daratumumab, and a glucocorticoid. There is no upper limit on the number of prior therapies provided that all other inclusion/exclusion criteria are met.
   * MM refractory to previous treatment with one or more glucocorticoids, parenteral PI (i.e., bortezomib and/or carfilzomib), IMiD (i.e., lenalidomide and/or pomalidomide), and the anti-CD38 mAb, daratumumab. Refractory is defined as ≤ 25% response to therapy, or progression during therapy or progression within 60 days after completion of therapy.

Exclusion Criteria:

* Active smoldering MM.
* Active plasma cell leukemia.
* Documented systemic amyloid light chain amyloidosis.
* Active CNS MM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (36):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic (AZ), Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Jonnsson Comprehensive Cancer Center / University of Los Angeles, Los Angeles, California
  - Smilow Cancer Hospital, New Haven, Connecticut
  - University of Florida Health Cancer Center- Shands Cancer Center Hospital, Gainesville, Florida
  - Sylvester, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center Research Institute, Tampa, Florida
  - Emory University / Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Kaiser Permanente- Hawaii, Honolulu, Hawaii
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Hackensack University Medical Center / John Therurer Cancer Center, Hackensack, New Jersey
  - Valley Hospital, Paramus, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Perlmutter Cancer Center, New York, New York
  - Mt Sinai NYC, New York, New York
  - Columbia University, New York, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Kaiser Permanente Northwest OR, Portland, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Ingram Cancer Center, Nashville, Tennessee
  - Baylor Sammons Cancer Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Austria (3):
  - University Hospital Krems, Department of Internal Medicine II, Krems
  - Salzburg Regional Hospital Müllner, Salzburg
  - Medical University Vienna, Department of Internal Medicine I, Vienna
- Belgium (7):
  - ZNA Stuivenberg, Antwerp
  - General Hospital Saint-Jan, Bruges
  - Jules Bordet Institute, Brussels
  - UCL Saint-Luc, Brussels
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Campus Gasthuisberg, Leuven
  - UCL Mont-Godinne, Yvoir
- France (7):
  - Claude Huriez Hospital, Department of Blood Diseases, Lille
  - South Lyon Hospital Center, Department of Clinical Hematology, Lyon
  - Brabois Adults Hospital, Nancy
  - Nantes University Hospital Center, Nantes
  - Hopital Saint-Antoine, Service d´Hematologie Clinique et Therapie Cellulaire, Paris
  - La Pitie-Salpetriere University Hospital, Department of Clinical Hematology, Paris
  - Necker Children's Hospital, Paris
- Germany (7):
  - BAG Oncology Gemeinschaftspraxis, Dresden
  - University Hospital Freiburg, Department of Internal Medicine I, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg Medizinische Klinik V, Heidelberg
  - Universitätsklinikum des Saarlandes Klinik für Innere Medizin I, Homburg
  - Universitätsmedizin Mainz, Mainz
  - University hospital of Tuebingen, Internal Medicine II, Tübingen
  - Med. Klinik und Poliklinik II Universitätsklinikum, Würzburg
- National & Kapodistrain University of Athens School of Medicine, Alexandra Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tremblay G, Daniele P, Breeze J, Li L, Shah J, Shacham S, Kauffman M, Engelhardt M, Chari A, Nooka A, Vogl D, Gavriatopoulou M, Dimopoulos MA, Richardson P, Biran N, Siegel D, Vlummens P, Doyen C, Facon T, Mohty M, Meuleman N, Levy M, Costa L, Hoffman JE, Delforge M, Kaminetzky D, Weisel K, Raab M, Dingli D, Tuchman S, Laurent F, Vij R, Schiller G, Moreau P, Richter J, Schreder M, Podar K, Parker T, Cornell RF, Lionel K, Choquet S, Sundar J. Quality of life analyses in patients with multiple myeloma: results from the Selinexor (KPT-330) Treatment of Refractory Myeloma (STORM) phase 2b study. BMC Cancer. 2021 Sep 6;21(1):993. doi: 10.1186/s12885-021-08453-9. PMID 34488662
- [Derived] Nikolaou A, Ambavane A, Shah A, Ma W, Tosh J, Kapetanakis V, Willson J, Wang F, Hogea C, Gorsh B, Gutierrez B, Sapra S, Suvannasankha A, Samyshkin Y. Belantamab mafodotin for the treatment of relapsed/refractory multiple myeloma in heavily pretreated patients: a US cost-effectiveness analysis. Expert Rev Hematol. 2021 Dec;14(12):1137-1145. doi: 10.1080/17474086.2021.1970522. Epub 2021 Sep 20. PMID 34465265
- [Derived] Chari A, Florendo E, Mancia IS, Cho H, Madduri D, Parekh S, Richter J, Dhadwal A, Thomas J, Jiang G, Lagana A, Bhalla S, Jagannath S. Optimal Supportive Care With Selinexor Improves Outcomes in Patients With Relapsed/Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2021 Dec;21(12):e975-e984. doi: 10.1016/j.clml.2021.07.014. Epub 2021 Jul 18. PMID 34404623
- [Derived] Chari A, Vogl DT, Gavriatopoulou M, Nooka AK, Yee AJ, Huff CA, Moreau P, Dingli D, Cole C, Lonial S, Dimopoulos M, Stewart AK, Richter J, Vij R, Tuchman S, Raab MS, Weisel KC, Delforge M, Cornell RF, Kaminetzky D, Hoffman JE, Costa LJ, Parker TL, Levy M, Schreder M, Meuleman N, Frenzel L, Mohty M, Choquet S, Schiller G, Comenzo RL, Engelhardt M, Illmer T, Vlummens P, Doyen C, Facon T, Karlin L, Perrot A, Podar K, Kauffman MG, Shacham S, Li L, Tang S, Picklesimer C, Saint-Martin JR, Crochiere M, Chang H, Parekh S, Landesman Y, Shah J, Richardson PG, Jagannath S. Oral Selinexor-Dexamethasone for Triple-Class Refractory Multiple Myeloma. N Engl J Med. 2019 Aug 22;381(8):727-738. doi: 10.1056/NEJMoa1903455. PMID 31433920
- [Derived] Vogl DT, Dingli D, Cornell RF, Huff CA, Jagannath S, Bhutani D, Zonder J, Baz R, Nooka A, Richter J, Cole C, Vij R, Jakubowiak A, Abonour R, Schiller G, Parker TL, Costa LJ, Kaminetzky D, Hoffman JE, Yee AJ, Chari A, Siegel D, Fonseca R, Van Wier S, Ahmann G, Lopez I, Kauffman M, Shacham S, Saint-Martin JR, Picklesimer CD, Choe-Juliak C, Stewart AK. Selective Inhibition of Nuclear Export With Oral Selinexor for Treatment of Relapsed or Refractory Multiple Myeloma. J Clin Oncol. 2018 Mar 20;36(9):859-866. doi: 10.1200/JCO.2017.75.5207. Epub 2018 Jan 30. PMID 29381435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 of the study was conducted at 32 sites in the United States and Part 2 of the study was conducted at 59 sites in France, Germany, Belgium, Greece, Austria and United States. Enrollment in both parts was between from 26 May 2015 (first participant first visit)) and 26 July 2019 (last participant last visit).
Pre-assignment Details: A total of 202 participants were enrolled in the study, out of which 79 participants were treated in Part 1 and 123 participants were treated in Part 2.
Period: Overall Study
Arm/Group | Part 1 | Part 2
Started | 79 | 123
Completed | 0 | 0
Not Completed | 79 | 123
Not completed — Disease Progression | 45 | 70
Not completed — Adverse Event | 18 | 39
Not completed — Physician Decision | 11 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other | 1 | 5

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants, who had received at least 1 dose of study treatment (partial or complete) and had any post-baseline safety information.
Groups:
- Part 1: Participants with quad-exposed, double-class-refractory (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, but not an anti-CD38 mab) and penta-exposed, triple-class-refractory MM (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, and daratumumab, and refractory to prior treatment with glucocorticoids, an IMiD, a PI, and the anti-CD38 mAb daratumumab) received, two dosing schedules (1) selinexor 80 mg plus low-dose dexamethasone 20 mg (Sd) twice-weekly on Days 1 and 3 for 3 weeks of each 4-week cycle (2) selinexor 80 mg plus low-dose dexamethasone 20 mg (Sd) twice-weekly continuously in 4-week cycles; until disease progression, death, or unacceptable toxicity (maximum duration of approximately 13 months).
- Part 2: Participants who previously had received more than 3 anti-MM regimens and had penta-exposed, triple class-refractory MM (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, and daratumumab, and refractory to prior treatment with glucocorticoids, an IMiD, a PI, and the anti-CD38 mAb daratumumab) received, selinexor 80 mg PO plus low-dose dexamethasone 20 mg Sd twice-weekly on Days 1 and 3 until disease progression, death, or unacceptable toxicity (maximum duration of approximately 17 months).
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 79 | 123 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.79) | 64.5 (9.41) | 63.9 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 52 | 94
  Male | 37 | 71 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 75 | 97 | 172
  Unknown or Not Reported | 2 | 17 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 21 | 35
  White | 62 | 86 | 148
  More than one race | 2 | 8 | 10
  Unknown or Not Reported | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Percentage of Participants With Overall Response Rate (ORR) Per International MyelomaWorking Group (IMWG) as Assessed by an Independent Review Committee (IRC)
Description: IRC assessed ORR per 2016 IMWG criteria: Percentage of participants who experienced Partial response (PR): greater than or equal to (>=) 50 percent (%) reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to lesser than (<) 200 mg per 24 hours; Very good partial response (VGPR): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours; Complete response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and lesser than or equal to (<=) 5% plasma cells in bone marrow; or stringent complete response (sCR): CR as defined+Normal free light chain (FLC) ratio+Absence of clonal cells in bone marrow biopsy by immunohistochemistry).
Time Frame: Baseline until disease progression/discontinuation from the study, or death, whichever occurred first (maximum duration of 17 months)
Population: Modified intent-to-treat (mITT) population consisted of Part 2 participants with penta-refractory MM who met all eligibility criteria and received at least one dose of study treatment. Data was not planned to be collected and analyzed for Part 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2
Number analyzed (Participants) | 122
Percentage of Participants | 26.2 [18.7 to 35.0]

2. Secondary Outcome: Part 1: Duration of Response (DoR) Per IMWG as Assessed by IRC
Description: IRC assessed DoR per 2016 IMWG criteria: time (in months) from the first documentation of objective response (confirmed CR or PR) to the date of first documentation of progressive disease (PD) or death due to any cause. Partial response (PR): >= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; Complete response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; Progressive disease (PD): Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 gram per deciliter (g/dL); Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urine M-protein (absolute increase must be >= 200 mg per 24 hours). Analysis was performed using Kaplan-Meier method.
Time Frame: First response subsequently confirmed to disease progression/discontinuation from the study, or death, whichever occurred first (maximum duration of 13 months)
Population: Safety population consisted of all participants, who had received at least 1 dose of study treatment (partial or complete) and had any post-baseline safety information. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1
Number analyzed (Participants) | 16
Months | 6.2 [3.6 to 9.8]

3. Secondary Outcome: Part 2: Duration of Response (DoR) Per IMWG as Assessed by an IRC
Description: IRC assessed DoR per 2016 IMWG criteria: time (in months) from the first documentation of objective response (confirmed CR or PR) to the date of first documentation of progressive disease (PD) or death due to any cause. Partial response (PR): >= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; Complete response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; Progressive disease (PD): Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >= 5 g/dL; Urine M-protein (absolute increase must be >= 200 mg per 24 hours). Analysis was performed using Kaplan-Meier method.
Time Frame: First response subsequently confirmed to disease progression/discontinuation from the study, or death, whichever occurred first (maximum duration of 17 months)
Population: mITT population consisted of Part 2 participants with penta-refractory MM who met all eligibility criteria and received at least one dose of study treatment. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2
Number analyzed (Participants) | 32
Months | 4.4 [3.7 to 10.8]

4. Secondary Outcome: Part 1: Percentage of Participants With Clinical Benefit Rate (CBR) ) Per IMWG as Assessed by IRC
Description: IRC assessed CBR per 2016 IMWG criteria: Percentage of participants with a confirmed minimal response (MR) or better (PR, VGPR, CR or sCR) before confirmed disease progression or initiating new MM treatment. Minimal response (MR): >= 25% but < 49% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 50-89%. Partial response (PR): >= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; Very good partial response (VGPR): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours; Complete response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; or stringent complete response (sCR): CR as defined+Normal free light chain (FLC) ratio+Absence of clonal cells by immunohistochemistry).
Time Frame: Baseline up to a maximum of 13 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1
Number analyzed (Participants) | 79
Percentage of Participants | 31.6 [21.6 to 43.1]

5. Secondary Outcome: Part 2: Percentage of Participants With Clinical Benefit Rate (CBR) Per IMWG as Assessed by IRC
Description: as for outcome 4
Time Frame: Baseline up to a maximum of 17 months
Population: mITT population consisted of Part 2 participants with penta-refractory MM who met all eligibility criteria and received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2
Number analyzed (Participants) | 122
Percentage of Participants | 39.3 [30.6 to 48.6]

6. Secondary Outcome: Part 1: Duration of Clinical Benefit Per IMWG as Assessed by IRC
Description: IRC assessed duration of clinical benefit per 2016 IMWG criteria: Duration from first response (at least MR) to time of IRC-determined PD or death due to disease progression, whichever occurs first. Minimal response (MR): >= 25% but < 49% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 50-89%. Progressive disease (PD): Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 hours). Analysis was performed using Kaplan-Meier method.
Time Frame: First response subsequently confirmed to disease progression, or death, whichever occurred first (maximum duration of 13 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1
Number analyzed (Participants) | 25
Months | 5.6 [4.4 to 10.3]

7. Secondary Outcome: Part 2: Duration of Clinical Benefit Per IMWG as Assessed by IRC
Description: as for outcome 6
Time Frame: First response subsequently confirmed to disease progression, or death, whichever occurred first (maximum duration of 17 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2
Number analyzed (Participants) | 48
Months | 3.8 [3.2 to 10.9]

8. Secondary Outcome: Part 2: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved stable disease (SD) or better (MR, PR, VGPR, CR, sCR) for a minimum of 12 weeks. Stable disease (SD): Not recommended for use as an indicator of response; stability of disease was best described by providing the time to progression (TTP) estimates. MR: >= 25% but < 49% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 50-89%. PR: >=50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <= 5% plasma cells in bone marrow; or sCR: CR as defined+Normal FLC ratio+Absence of clonal cells by immunohistochemistry).
Time Frame: Every 12 weeks until progressive disease or death due to any cause, up to 17 months
Population: mITT population consisted of Part 2 participants with penta-refractory MM who met all eligibility criteria and received at least one dose of study treatment. Data was not planned to be collected and analyzed for Part 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2
Number analyzed (Participants) | 122
Percentage of Participants | 44.3 [35.3 to 53.5]

9. Secondary Outcome: Part 1: Progression Free Survival (PFS) Per IMWG as Assessed by IRC
Description: IRC assessed PFS per 2016 IMWG criteria: Duration from start of study treatment until IRC-determined progressive disease (PD) or death from any cause, whichever occurred first. Progressive disease (PD): Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >=1 g/dL if the lowest M-component was >= 5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg/24 hours). Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment to progression of disease or discontinuation from the study or death, whichever occurred first (maximum duration of 13 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1
Number analyzed (Participants) | 79
Months | 4.7 [3.3 to 7.6]

10. Secondary Outcome: Part 2: Progression Free Survival (PFS) Per IMWG as Assessed by IRC
Description: as for outcome 9
Time Frame: From start of study treatment to progression of disease or discontinuation from the study or death, whichever occurred first (maximum duration of 17 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2
Number analyzed (Participants) | 122
Months | 3.7 [2.8 to 4.7]

11. Secondary Outcome: Part 1: Time to Progression (TTP) Per IMWG as Assessed by IRC
Description: IRC assessed TTP per 2016 IMWG criteria: Duration from start of study treatment until PD or death due to PD (per IRC), whichever occurred first. Progressive disease (PD): Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >=1 g/dL if the lowest M-component was >= 5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg/24 hours). Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment to progression of disease or death, whichever occurred first (maximum duration of 13 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1
Number analyzed (Participants) | 79
Months | 5.5 [3.3 to 10.7]

12. Secondary Outcome: Part 2: Time to Progression (TTP) Per IMWG as Assessed by IRC
Description: as for outcome 11
Time Frame: From start of study treatment to progression of disease or death, whichever occurred first (maximum duration of 17 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2
Number analyzed (Participants) | 122
Months | 4.1 [3.0 to 6.2]

13. Secondary Outcome: Part 1: Time to Next Treatment (TTNT)
Description: TTNT was defined as the duration from start of study treatment to start of next anti-MM treatment or death due to disease progression, whichever occurred first. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment to start of next anti-MM treatment or death due to disease progression, whichever occurs first (maximum duration of 13 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1
Number analyzed (Participants) | 79
Months | 2.6 [1.8 to 4.2]

14. Secondary Outcome: Part 2: Time to Next Treatment (TTNT)
Description: as for outcome 13
Time Frame: From start of study treatment to start of next anti-MM treatment or death due to disease progression, whichever occurs first (maximum duration of 17 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2
Number analyzed (Participants) | 122
Months | 3.2 [2.6 to 3.8]

15. Secondary Outcome: Part 1: Overall Survival (OS)
Description: OS was defined as the duration (in months) from start of study treatment to death from any cause. Participants last known to be alive were censored at the date of discontinuation from the study, or database cut date, whichever was earlier. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment to death (maximum duration of 13 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1
Number analyzed (Participants) | 79
Months | 7.3 [5.8 to 10.9]

16. Secondary Outcome: Part 2: Overall Survival (OS)
Description: as for outcome 15
Time Frame: From start of study treatment to death (maximum duration of 17 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2
Number analyzed (Participants) | 122
Months | 8.4 [6.2 to 11.2]

17. Secondary Outcome: Part 2: Change From Baseline in Health-related Quality of Life (HRQL) Score Based on Functional Assessment of Cancer Therapy - Multiple Myeloma (FACT-MM) Questionnaire
Description: FACT-MM combines the general version of the FACT (FACT-G) with a MM-specific sub-scale (14 items). The sub-scales for the FACT-G are Physical Well-Being (7 items), Social/Family Well-Being (7 items), Emotional Well-Being (6 items), and Functional Well-Being (7 items). The trial outcomes index (TOI); total of 41 items) is the primary measurement of interest, comprised of the Physical and Functional sub-scales plus the MM-specific sub-scale. Each item is rated on a 5-point Likert scale, ranging from 0 ("Not at all") to 4 ("Very much"), therefore the TOI has a score ranging from 0 to 120. Higher scores indicated improvement in well being.
Time Frame: Baseline, Day 1 of Cycle 2 to Cycle 20 (up to a maximum of 17 months)
Population: mITT population set. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure at given time points. Data was not planned to be collected and analyzed for Part 1.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part 2
Number analyzed (Participants) | 107
Score on a Scale
  Trial Outcomes Index Score: Baseline | 67.5 (19.20)
  Trial Outcomes Index Score: Change at C2D1: number analyzed (Participants) | 76
  Trial Outcomes Index Score: Change at C2D1 | -6.1 (18.43)
  Trial Outcomes Index Score: Change at C3D1: number analyzed (Participants) | 50
  Trial Outcomes Index Score: Change at C3D1 | -8.5 (15.50)
  Trial Outcomes Index Score: Change at C4D1: number analyzed (Participants) | 31
  Trial Outcomes Index Score: Change at C4D1 | -9.1 (16.79)
  Trial Outcomes Index Score: Change at C5D1: number analyzed (Participants) | 26
  Trial Outcomes Index Score: Change at C5D1 | -6.9 (12.06)
  Trial Outcomes Index Score: Change at C6D1: number analyzed (Participants) | 19
  Trial Outcomes Index Score: Change at C6D1 | -8.3 (15.07)
  Trial Outcomes Index Score: Change at C7D1: number analyzed (Participants) | 13
  Trial Outcomes Index Score: Change at C7D1 | -7.5 (19.26)
  Trial Outcomes Index Score: Change at C8D1: number analyzed (Participants) | 5
  Trial Outcomes Index Score: Change at C8D1 | -15.4 (24.59)
  Trial Outcomes Index Score: Change at C9D1: number analyzed (Participants) | 3
  Trial Outcomes Index Score: Change at C9D1 | -4.7 (14.84)
  Trial Outcomes Index Score: Change at C10D1: number analyzed (Participants) | 3
  Trial Outcomes Index Score: Change at C10D1 | -4.0 (5.29)
  Trial Outcomes Index Score: Change at C11D1: number analyzed (Participants) | 1
  Trial Outcomes Index Score: Change at C11D1 | 3.0 (NA) — Standard deviation was not estimated due to single participant.
  Trial Outcomes Index Score: Change at C12D1: number analyzed (Participants) | 1
  Trial Outcomes Index Score: Change at C12D1 | 3.0 (NA) — Standard deviation was not estimated due to single participant.
  Trial Outcomes Index Score: Change at C13D1: number analyzed (Participants) | 1
  Trial Outcomes Index Score: Change at C13D1 | -23.0 (NA) — Standard deviation was not estimated due to single participant.
  Trial Outcomes Index Score: Change at C14D1: number analyzed (Participants) | 1
  Trial Outcomes Index Score: Change at C14D1 | 14.0 (NA) — Standard deviation was not estimated due to single participant.
  Trial Outcomes Index Score: Change at C15D1: number analyzed (Participants) | 1
  Trial Outcomes Index Score: Change at C15D1 | 1.0 (NA) — Standard deviation was not estimated due to single participant.
  Trial Outcomes Index Score: Change at C16D1: number analyzed (Participants) | 1
  Trial Outcomes Index Score: Change at C16D1 | 4.0 (NA) — Standard deviation was not estimated due to single participant.
  Trial Outcomes Index Score: Change at C17D1: number analyzed (Participants) | 0
  Trial Outcomes Index Score: Change at C18D1: number analyzed (Participants) | 0
  Trial Outcomes Index Score: Change at C19D1: number analyzed (Participants) | 0
  Trial Outcomes Index Score: Change at C20D1: number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) of Grade 3/4, Graded Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Treatment-emergent events are events between first dose of study drug and up to last dose of study treatment + 30 days (inclusive) that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline to 30 days after last dose of study treatment (maximum duration of 18 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 79 | 123
Participants | 75 | 115

19. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (TEAEs) of Grade 3/4, Graded Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. A treatment related AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event had a causal relationship with the treatment or usage.
Time Frame: Baseline to 30 days after last dose of study treatment (maximum duration of 18 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Participants with quad-exposed, double-class-refractory (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, but not an anti-CD38 mab) and penta-exposed, triple-class-refractory MM (i.e. previously treated with lenalidomide, pomalidomide, bortezomib, carfilzomib, and daratumumab, and refractory to prior treatment with glucocorticoids, an IMiD, a PI, and the anti-CD38 mAb daratumumab) received, two dosing schedules (1) selinexor 80 mg plus low-dose dexamethasone 20 mg (Sd) twice-weekly on Days 1 and 3 for 3 weeks of each 4-week cycle (2) selinexor 80 mg plus low-dose dexamethasone 20 mg (Sd) twice-weekly continuously in 4-week cycles; until disease progression, death, or unacceptable toxicity (maximum duration of approximately 13 months
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 79 | 123
Participants | 69 | 110

20. Secondary Outcome: Apparent Clearance (CL/F) of Selinexor in Plasma
Description: CL/F of selinexor in plasma was reported.
Time Frame: Cycle 1: Day 1: Pre-dose, 1, 2 and 4 hours post-dose; Day 8 and 15: Pre-dose and 1 hour post-dose; Cycle 2: Day 1: Predose, 1, 2 and 4 hours post-dose
Population: Pharmacokinetic (PK) set included all participants in Part 1 who received at least 1 dose of investigational product in this study. Data was not planned to be collected and analyzed for Part 2.
Measure: Mean (Standard Deviation); unit: Liters/Hour
Arm/Group | Part 1
Number analyzed (Participants) | 79
Liters/Hour | 16.6 (2.8)

21. Secondary Outcome: Volume of Distribution (V/F) of Selinexor in Plasma
Description: Vz/F of selinexor in plasma was reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part 1
Number analyzed (Participants) | 79
Liter | 145.6 (28.2)

ADVERSE EVENTS:
Time Frame: Baseline to 30 days after last dose of study treatment (maximum duration of 18 months)
Arm/Group | Part 1 | Part 2
All-Cause Mortality (participants affected / at risk) | 20/79 | 28/123
Serious Adverse Events (participants affected / at risk) | 45/79 | 78/123
Other Adverse Events (participants affected / at risk) | 79/79 | 123/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (N=79) | Part 2 (N=123)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Asthenia (General disorders) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 14 (14)
Sepsis (Infections and infestations) | 1 (1) | 12 (12)
Bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Respiratory syncytial virus test positive (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 4 (4)
Mental status changes (Psychiatric disorders) | 1 (1) | 4 (4)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Strangulated hernia (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (N=79) | Part 2 (N=123)
Thrombocytopenia (Blood and lymphatic system disorders) | 58 (58) | 91 (91)
Anaemia (Blood and lymphatic system disorders) | 37 (37) | 80 (80)
Neutropenia (Blood and lymphatic system disorders) | 23 (23) | 49 (49)
Leukopenia (Blood and lymphatic system disorders) | 20 (20) | 41 (41)
Lymphopenia (Blood and lymphatic system disorders) | 11 (11) | 20 (20)
Tachycardia (Cardiac disorders) | 9 (9) | 4 (4)
Vision blurred (Eye disorders) | 10 (10) | 13 (13)
Nausea (Gastrointestinal disorders) | 60 (60) | 88 (88)
Diarrhoea (Gastrointestinal disorders) | 35 (35) | 57 (57)
Vomiting (Gastrointestinal disorders) | 37 (37) | 47 (47)
Constipation (Gastrointestinal disorders) | 21 (21) | 27 (27)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 12 (12)
Fatigue (General disorders) | 55 (55) | 77 (77)
Pyrexia (General disorders) | 10 (10) | 18 (18)
Asthenia (General disorders) | 5 (5) | 19 (19)
Oedema peripheral (General disorders) | 5 (5) | 14 (14)
Chills (General disorders) | 6 (6) | 4 (4)
Malaise (General disorders) | 2 (2) | 8 (8)
Gait disturbance (General disorders) | 0 (0) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 17 (17)
Pneumonia (Infections and infestations) | 3 (3) | 10 (10)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 13 (13)
Weight decreased (Investigations) | 39 (39) | 61 (61)
Alanine aminotransferase increased (Investigations) | 6 (6) | 13 (13)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 11 (11)
Decreased appetite (Metabolism and nutrition disorders) | 43 (43) | 68 (68)
Hyponatraemia (Metabolism and nutrition disorders) | 34 (34) | 45 (45)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (16) | 15 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 24 (24)
Dehydration (Metabolism and nutrition disorders) | 15 (15) | 10 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 13 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (10) | 10 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 8 (8)
Hypercreatininaemia (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (11)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 12 (12) | 19 (19)
Headache (Nervous system disorders) | 10 (10) | 11 (11)
Dysgeusia (Nervous system disorders) | 10 (10) | 10 (10)
Peripheral neuropathy (Nervous system disorders) | 7 (7) | 8 (8)
Insomnia (Psychiatric disorders) | 11 (11) | 22 (22)
Confusional state (Psychiatric disorders) | 9 (9) | 11 (11)
Anxiety (Psychiatric disorders) | 4 (4) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 28 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 18 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 13 (13)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02336815/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT02336815/SAP_001.pdf